CLINICAL TRIAL: NCT06561373
Title: Mindfulness-Based Intervention: Effects on Emotional Regulation, Behavior, and Social Participation for Preschool Students
Brief Title: Effects of Mindfulness and Yoga on Preschool Students' Emotional Regulation, Behavior, and Social Participation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Elizabethtown College (Other)
Responsible Party: Principal Investigator, Helen Russell, Dr. Helen Russell, pp-OTD, Elizabethtown College
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2185448-1
Record Dates: First submitted 2024-08-16; First posted 2024-08-20 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Prosocial Behavior; Self Regulation; Impulsive Behavior
Keywords: mindfulness; children; yoga; preschool; school-based intervention; self-regulation; behavioral incident; occupational therapy
MeSH Terms: conditions — Altruism; Self-Control; Impulsive Behavior | interventions — Calmodulin; Mindfulness; Yoga

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The secondary researchers will be blinded to which students are in the control and intervention groups until after they have run the statistical analyses.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Calm and Alert Mindfulness and Yoga Intervention (Experimental): The Calm & Alert intervention uses mind, body, and breath to foster resiliency and self-regulation in students. This mindfulness-based intervention, which also incorporates yoga movements, aims to develop skills in self-awareness, self-regulation, safety, focus, attention, active listening, following directions, respect, and positive thinking (McGlauflin, 2018). The program consisted of seven lessons lasting approximately 20-30 minutes, each conducted once a week over seven consecutive weeks.
  Interventions: Behavioral: Calm & Alert yoga and mindfulness
- Control Group (No Intervention): This is a wait-list control group that consists of students in classrooms who will receive business-as-usual programming/instruction during the study period.

INTERVENTIONS:
Behavioral: Calm & Alert yoga and mindfulness — The Calm & Alert protocol is multisensorial, with successive opportunities to practice the explicit concepts taught throughout the lessons using yoga and mindfulness-techniques. Each class has a similar structure of songs, breathing, warm-ups, yoga poses, mindful games, and rest involving meditation with child-friendly language. The study includes the recommended materials of a Hoberman sphere (breathing ball), chime, mind/body/breath icons, two small mason jars (one with mud and one with clear water), yoga mats for students, pictures of feelings (happy, sad, angry, scared, surprised, disgusted), and an on/off switch.
  Other Names: yoga and mindfulness; mindfulness-based intervention
  Arms: Calm and Alert Mindfulness and Yoga Intervention

SUMMARY:
The goal of this clinical trial is to learn if mindfulness and yoga can improve attention, problem-solving, memory, emotional awareness, and impulsivity in preschoolers. The main questions it aims to answer are:

Can a 30-minute, once-a-week mindfulness and yoga program (Calm & Alert) over seven weeks in preschool classrooms increase emotional regulation during the school day? Can a 30-minute, once-a-week mindfulness and yoga program decrease negative behavioral incidences during the school day? Can a 30-minute, once-a-week mindfulness and yoga program increase prosocial behaviors like caring, sharing, and perspective-taking during the school day? Researchers will compare the effects of students who participated in the mindfulness and yoga program to students in classrooms who did not receive the program. Student participants will be asked to complete a short self-regulation task test before and after the mindfulness program. Teachers will rate the students on their prosocial behavior before and after the mindfulness program and record negative behavioral incidents over the study period.

DETAILED DESCRIPTION:
The current study design is a quasi-experimental pretest post-study design with a control group. Three schools with a total of four preschool classrooms will participate in this study. Overall, the present research study aims to add to the knowledge base of the benefits of mindfulness and yoga in schools for young children. This will include investigating the effect of mindfulness on children's attention, problem-solving, memory, emotional awareness, and impulsivity. For seven weeks, the intervention group will receive the Calm & Alert mindfulness intervention alongside the rest of their class involving one session per week of about 30 minutes of yoga and mindfulness. The control group will conduct business as usual and receive the yoga and mindfulness intervention after the study concludes. The intervention will be provided by the principal investigator who is a certified mindfulness-informed professional and registered yoga teacher - 200 hours. It is hypothesized that implementing a 30-minute, once-a-week mindfulness program over seven weeks in preschool classrooms will increase emotional regulation, decrease negative behavioral incidents, and increase prosocial behaviors during the school day.

ELIGIBILITY:
Inclusion Criteria:

* are preschoolers with a filled out and returned parental/caregiver consent form who fall within the four to six-year-old age range, stay within a similar developmental age range, and attend five out of the seven sessions.

Exclusion Criteria: preschoolers without a parental/caregiver consent form, above or below the four to six-year age range will not be included in the study because of the higher variation in developmental capabilities, and if they do not attend five out of the seven sessions.

-

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2024-08-23 (Estimated); Primary Completion 2024-11-11 (Estimated); Study Completion 2024-11-11 (Estimated)

PRIMARY OUTCOMES:
Strengths and Difficulties Questionnaire | Pre-intervention and post-intervention (within one week)
  The Strengths and Difficulties Questionnaire - Teacher Form (SDQ) is a widely used behavioral screening questionnaire that correlates highly with measures of behavior problems (Goodman & Scott, 1999). The teacher form asks teachers to rate classroom students according to their perceived behavior. It consists of 25 items divided into five scales: emotional symptoms, conduct problems, hyperactivity/inattention, peer relationship problems, and prosocial behavior. For this study, the prosocial behavior subscale will be primarily used for pre- and post-assessment data analysis. The teacher form asks teachers to rate classroom students according to their perceived behavior.
Head-Toes-Knees-Shoulders Task | Pre-intervention and post-intervention (within one week for post and before the start of the study period for pretest)
  The Head-Toes-Knees-Shoulders (HTKS) Task is an ecologically valid method to measure behavioral aspects of self-regulation, such as controlling and directing actions, inhibitory control, paying attention, and recalling instructions (Ponitz, 2008; McClelland and Cameron, 2012). The test is introduced as a game with a gross motor component that more closely aligns with self-regulation behaviors required of children within natural contexts such as the classroom (McClelland and Cameron, 2012).

SECONDARY OUTCOMES:
Negative Behavior Incidents | during the intervention period.
  School teachers will track behavioral incidents that fall outside the expected behavior realm for student participants.

CONTACTS AND LOCATIONS:
Overall Officials: Helen C Russell, doctorate, Principal Investigator — Elizabethtown College; Ella Longenecker, Bachelor, Study Chair — Elizabethtown College; Samantha Deiaco, Bachelor, Study Chair — Elizabethtown College; Ellysa Herr, Bachelor, Study Chair — Elizabethtown College; Sarah Lloyd, Bachelor, Study Chair — Elizabethtown College
Locations (1):
- Elizabethtown College, Elizabethtown, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Identifying information of the minors that are study participants will not be shared.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: anticipated within 6 months of study completion
Access Criteria: Per request

REFERENCES:
- [Background] Carro N, D'Adamo P, Lozada M. A School Intervention Helps Decrease Daily Stress While Enhancing Social Integration in Children. Behav Med. 2021 Jul-Sep;47(3):251-258. doi: 10.1080/08964289.2020.1738319. Epub 2020 Apr 10. PMID 32275198
- [Background] Goodman, R. (1997). Strengths and Difficulties Questionnaire (SDQ) [Database record]. APA PsycTests. https://doi.org/10.1037/t00540-000
- [Background] McClelland, M. M., Cameron, C., Bowles, R., & Geldhof, G. (2018). Developing a measure of self-regulation for at-risk children. U.S. Department of Education, Institute for Education Sciences.
- [Background] McGlauflin, H. (2018). Calm & Alert: Yoga and mindfulness practices to teach self-regulation and social skills to children (1st ed.). PESI Publishing & Media.
- [Background] Rashedi RN, Rowe SE, Thompson RA, Solari EJ, Schonert-Reichl KA. A Yoga Intervention for Young Children: Self-Regulation and Emotion Regulation. J Child Fam Stud. 2021;30(8):2028-2041. doi: 10.1007/s10826-021-01992-6. Epub 2021 Jun 9. PMID 34127901
- [Background] Sciutto MJ, Veres DA, Marinstein TL, Bailey BF, Cehelyk SK. Effects of a School-Based Mindfulness Program for Young Children. J Child Fam Stud. 2021;30(6):1516-1527. doi: 10.1007/s10826-021-01955-x. Epub 2021 Apr 15. PMID 33875914